CLINICAL TRIAL: NCT04120155
Title: Preservation vs. Dissection of Inferior Pulmonary Ligament for Thoracoscopic Upper Lobectomy: A Prospective Randomized Controlled Trial（IPLP FJUNION）
Brief Title: Preservation vs. Dissection of Inferior Pulmonary Ligament for Thoracoscopic Upper Lobectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Collaborators: Fuqing City Hospital (Unknown); Sanming Second Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPLP FJUNION
Record Dates: First submitted 2019-09-18; First posted 2019-10-09 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dissecting the inferior pulmonary ligament (Other): This group of patients will undergo the inferior pulmonary dessection during the upper lobe thoractomy.
  Interventions: Procedure: Dissection of the Inferior Pulmonary Ligament
- Preserving the inferior pulmonary ligament (Other): This group of patients will undergo the inferior pulmonary preservation during the upper lobe thoractomy.
  Interventions: Procedure: Preservation of the Inferior Pulmonary Ligament

INTERVENTIONS:
Procedure: Dissection of the Inferior Pulmonary Ligament — Patients will be categorized into two groups: the division group ,who will receive the division of the inferior pulmonary ligament, and the preservation group, who will not.For the dissection group, we will dissect the inferior pulmonary ligament during the surgery.
  Arms: Dissecting the inferior pulmonary ligament
Procedure: Preservation of the Inferior Pulmonary Ligament — Patients will be categorized into two groups: the division group ,who will receive the division of the inferior pulmonary ligament, and the preservation group, who will not.For the preservation group, we will preserve the inferior pulmonay ligament during the surgery.
  Arms: Preserving the inferior pulmonary ligament

SUMMARY:
Many thoracic surgeons tend to dissect the inferior pulmonary ligament (IPL) during upper lobectomy, which in theory reduces the free space in the upper thoracic cavity by increasing the mobility of the residual lung. However, the dissection of IPL may lead to bronchial deformation, stenosis, obstruction or lobe torsion, and distortion. Some studies have found that stenosis might be associated with chronic dry cough and shortness of breath, and could result in a significant decline in lung function. Moreover, the dissection of IPL may lead to greater surgical trauma and increase the incidence of complications. Therefore, this study tries to identify whether we should dissect or preserve the inferior pulmonary ligament during the thoracoscopic upper lobectomy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old < age < 70 years old;
2. Meet the indications for thoracoscopic left/right upper lobectomy;
3. Gave informed consent and were willing to undergo thoracoscopic left/right upper lobectomy;
4. Preoperative pulmonary function test: FEV1>1L and FEV1>60% of the predicted value;
5. Preoperative ECOG score of 0-1;
6. Preoperative ASA score I-II.

Exclusion Criteria:

1. Inferior mediastinal lymphadenopathy was found in preoperative screening;
2. Found that other lobe operations were required at the same time due to multiple lesions in the preoperative discussion;
3. Pregnant or lactating women;
4. Suffering from severe mental illness;
5. History of thoracic surgery (including intrathoracic surgery only, excluding surface surgery such as mastectomy);
6. History of unstable angina or myocardial infarction within the past six months;
7. History of cerebral infarction or cerebral hemorrhage within the past six months;
8. History of continuous systemic corticosteroid therapy within the past month;
9. Abnormal coagulation function, bleeding tendency, or receiving antithrombotic or antiplatelet therapy recently;
10. Suffering from severe liver, kidney, and other systemic diseases;
11. Other situations that are not suitable for surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in bronchial angle | 3 months after the operation
  Change in bronchial angle of each arm(measured by coronal CT)
Change in bronchial angle | 6 months after the operation
  Change in bronchial angle of each arm(measured by coronal CT)
Change in lung volume | 3 months after the operation
  Change in lung volume of each arm(measured by Mimics Research 21.0 software)
Change in lung volume | 6 months after the operation
  Change in lung volume of each arm(measured by Mimics Research 21.0 software)

SECONDARY OUTCOMES:
Apical dead space | Within 6 months after the operation
  Apical dead space incidence rate
Pleural effusion | Within 6 months after the operation
  Pleural effusion incidence rate
Lung infection | Within 6 months after the operation
  Lung infection incidence rate
Atrial fibrillation | During the postoperative hospital stay
  Atrial fibrillation incidence rate
Operation time | During the operation
  Operation time
Postoperative hospital stay | During the postoperative hospital stay
  Postoperative hospital stay
Closed thoracic drainage tube rentention time | During the postoperative hospital stay
  Closed thoracic drainage tube rentention time
Disposable drainage catheter retention time | Within one month after the operation
  Disposable drainage catheter retention time
Pathologic cancer stage | After the operation
  Pathologic cancer stage
Histologic diagnosis | After the operation
  Histologic diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Chun Chen, MD, Study Director — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China